CLINICAL TRIAL: NCT03782675
Title: Air Barrier System for the Reduction of Airborne Particulate and Colony-forming Units (CFU) During Total Shoulder Arthroplasty.
Brief Title: Air Barrier System for the Reduction of Airborne Colony-forming Units During Total Shoulder Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nimbic Systems, LLC (Industry)
Collaborators: Texas Orthopedic Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: ABS-104
Record Dates: First submitted 2018-12-13; First posted 2018-12-20 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Osteo Arthritis Shoulders
Keywords: Total shoulder replacement; operating room air; surgical site infection; airborne CFU
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control (Sham Comparator): In the control arm, the ABS device will be placed as usual on the patient, but the airflow will NOT be activated. Only the technician in the room will be aware whether the device the device is turned on or not.
  Interventions: Device: Control
- Air Barrier System (Experimental): In the experimental (interventional) arm, the ABS device will be placed as usual on the patient, and the airflow will be activated. Only the technician in the room will be aware whether the device is turned on or not.
  Interventions: Device: Air Barrier System

INTERVENTIONS:
Device: Control — The Air Barrier System will be deployed onto the surgical field, but the airflow will not be activated, so this is a sham control comparator.
  Arms: Control
Device: Air Barrier System — The Air Barrier System is a device that uses localized clean air flow to shield a surgery site from ambient airborne microorganisms that are shed into the air from people present in the operating room.
  Arms: Air Barrier System

SUMMARY:
The objective of this study is to determine whether the Air Barrier System device reduces airborne colony-forming units (e.g., bacteria) present at a surgery site during total shoulder arthroplasty surgeries.

DETAILED DESCRIPTION:
The Air Barrier System (ABS) is a device that uses localized clean air flow to shield a surgery site from ambient airborne contamination. This study examines the hypothesis that the ABS can reduce the presence of airborne CFU and particles at the surgery site during total arthroplasty surgery.

ELIGIBILITY:
Inclusion Criteria:

* Candidate for total shoulder arthroplasty

Exclusion Criteria:

* Prior history of infection
* Revision surgery
* Screens positive for MRSA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-02 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
CFU counts | Four months
  Inter-arm comparison of CFU counts taken during both the Control arm and ABS arm
Particle counts | Four months
  Inter-arm comparison of particle counts taken during both the Control arm and ABS arm.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Stocks, MD, Principal Investigator — Texas Orthopedic Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stocks GW, Self SD, Thompson B, Adame XA, O'Connor DP. Predicting bacterial populations based on airborne particulates: a study performed in nonlaminar flow operating rooms during joint arthroplasty surgery. Am J Infect Control. 2010 Apr;38(3):199-204. doi: 10.1016/j.ajic.2009.07.006. Epub 2009 Nov 12. PMID 19913327